CLINICAL TRIAL: NCT00483353
Title: A Pilot Study to Explore the Effect of a Nasal Bolus Allergen Challenge on Inflammatory Markers in Subjects With Seasonal Allergic Rhinitis
Brief Title: Effect of a Nasal Bolus Allergen Challenge on Inflammatory Markers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9011058
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

INTERVENTIONS:
Procedure: Intra-nasal allergen challenge with Phleum pratense.
Procedure: Collection of nasal effluent using filter paper.
Procedure: Measurement of nasal congestion using acoustic rhinometry.

SUMMARY:
The current study will investigate nasal inflammatory markers obtained by filter paper collection techniques, in subjects with allergic rhinitis, determining the most appropriate time points and handling conditions, prior to running a larger study with subjects with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with allergic rhinitis, that have a positive skin prick response to Phleum pratense.

Exclusion Criteria:

* Subjects with a history of asthma. Current smokers, or recent ex-smokers and subjects that have had a respiratory tract infection in the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2007-07

PRIMARY OUTCOMES:
Post allergen challenge nasal inflammatory markers at 1, 5, 15, 30, 45 min, 1, 2, 3, 4, 5, 6, 7, 8 hours post allergen challenge.

SECONDARY OUTCOMES:
Post allergen challenge effects on acoustic rhinometry and symptoms at 16, 31, 45 min, 1, 2, 3, 4, 5, 6, 7, 8 hours post allergen challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, London, England, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011058&StudyName=Effect%20of%20a%20nasal%20bolus%20allergen%20challenge%20on%20inflammatory%20markers%20